CLINICAL TRIAL: NCT04663204
Title: A Multi-centre, Open-label, Single-group Exploratory Trial of the Safety and Activity of Sparsentan for the Treatment of Incident Patients With Immunoglobulin A Nephropathy
Brief Title: A Study of the Safety and Activity of Sparsentan for the Treatment of Incident Patients With Immunoglobulin A Nephropathy
Acronym: SPARTAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0708; 2018-002012-27 (EudraCT Number); 257450 (Other: Health Research Authority)
Record Dates: First submitted 2020-12-08; First posted 2020-12-10 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Immunoglobulin A Nephropathy; Kidney Diseases; Glomerulonephritis, IGA; Glomerulonephritis; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Glomerulonephritis; Autoimmune Diseases; Immune System Diseases | interventions — sparsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sparsentan (Experimental): Sparsentan will be administered once daily, starting at a dose of 200 mg (two 100 mg oral capsules) for the first 2 weeks of the study. Patients who tolerate the initial dose of 200 mg after 2 weeks will increase their dose to 400 mg (one 400 mg tablet). Patients who do not tolerate the target dose will have their dose reduced back to 200 or 100 mg/day; throughout the study, patients will be maintained on the maximum allowed dose of sparsentan they can tolerate. All patients will be treated with sparsentan for a total of 110 weeks.
  Interventions: Drug: Sparsentan

INTERVENTIONS:
Drug: Sparsentan — Target dose of 400 mg daily
  Other Names: RE-021

SUMMARY:
To determine the nephroprotective potential of treatment with sparsentan in patients newly-diagnosed with immunoglobulin A nephropathy (IgAN) (ie, incident patients) who have not received prior angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) therapy.

DETAILED DESCRIPTION:
A multi-centre, open-label, single-group trial is proposed to explore the safety of, and response to sparsentan treatment in incident, renin angiotensin system (RAS) blockade-naïve patients with biopsy-proven immunoglobulin A nephropathy (IgAN).

The purpose is to explore sparsentan treatment as a potential first-line treatment in patients newly diagnosed with IgAN (ie, incident patients), who have thus not received prior treatment with ACEI or ARB therapy for IgAN. Response to treatment will be assessed as changes from baseline rather than comparison to another treatment, and will be based on established proteinuria endpoints (UPCR and protein excretion), and glomerular filtration rate (GFR); a number of exploratory measures will be assessed as well.

The starting dose of sparsentan will be 200 mg/day, which will be titrated up to the target dose of 400 mg/day at Week 2. Patients who do not tolerate the target dose will have their dose reduced back to 200 or 100 mg/day; throughout the study, patients will be maintained on the maximum allowed dose of sparsentan they can tolerate. All patients will be treated with sparsentan for a total of 110 weeks, followed by an off-treatment follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to provide signed informed consent.
* The patient can understand written and spoken English.
* The patient is male or female, aged ≥18 years.
* The patient has been diagnosed with biopsy-proven IgAN within the last 6 months (calculated from the date of kidney biopsy, upon which the IgAN-positive diagnosis was made, to the signing of the informed consent form).
* The patient has a urine total protein value ≥0.5 g/day at screening.
* The patient has an eGFR value ≥30 mL/min/1.73 m2 at screening.
* The patient has not previously been treated with ACEI and/or ARB therapy for IgAN OR has not received ACEI and/or ARB therapy within the last 12 months.
* The patient has a systolic BP ≤150 mmHg and ≥100 mmHg, and diastolic blood pressure ≤100 mmHg and ≥60 mmHg at screening.
* Women of childbearing potential (WOCBP), beginning at menarche, must agree to the use of one highly reliable (ie, can achieve a failure rate of <1% per year) method of contraception from 7 days prior to the first dose of trial medication until 90 days after the last dose of trial medication. Highly reliable contraception methods include stable oral, implanted, transdermal, or injected contraceptive hormones associated with inhibition of ovulation, or an intrauterine device (IUD) in place for at least 3 months. One additional barrier method must also be used during sexual activity, such as a diaphragm or diaphragm with spermicide (preferred), or male partner's use of male condom or male condom with spermicide), from Day 1 until 90 days after the last dose of trial medication.

WOCBP are defined as those who are fertile, following menarche and until becoming postmenopausal unless permanently sterile; permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as amenorrhoea for more than 24 consecutive months without an alternative medical cause; women on hormone replacement therapy must have a documented plasma follicle-stimulating hormone level ≥40 mIU/mL. All WOCBP must have a negative pregnancy test at Visit 1 (serum test) and Visit 2 (urine, with positive results confirmed by serum).

Exclusion Criteria:

* The patient has IgAN secondary to another condition (eg, systemic lupus erythematosus, liver cirrhosis).
* The patient, in the opinion of the Investigator, has a rapidly progressive glomerulonephritis (rapid decline in GFR and crescents on biopsy).
* The patient has a history of type 1 diabetes mellitus, uncontrolled type 2 diabetes mellitus (haemoglobin A1c [HbA1c] >8%), or nonfasting blood glucose >10 mmol/L (180 mg/dL) at screening.
* The patient has undergone any organ transplantation, with the exception of corneal transplants.
* The patient requires any of the prohibited concomitant medications (see Section 14.4).
* The patient has been taking any systemic immunosuppressive medications for >2 weeks within 6 months prior to screening.
* The patient has a documented history of heart failure (New York Heart Association Class II-IV) and/or previous hospitalisation for heart failure or unexplained dyspnoea, orthopnoea, paroxysmal nocturnal dyspnoea, ascites, and/or peripheral oedema.
* The patient has clinically significant cerebrovascular disease (transient ischemic attack or stroke) and/or coronary artery disease (hospitalisation for myocardial infarction or unstable angina, new onset of angina with positive functional tests, coronary angiogram revealing stenosis, or a coronary revascularisation procedure) within 6 months prior to screening.
* The patient has jaundice, hepatitis, or known hepatobiliary disease (including asymptomatic cholelithiasis), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of the normal range at screening.
* The patient has a history of malignancy other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma within the past 2 years.
* The patient has a screening haematocrit value <27% or haemoglobin value <90 g/L (9 g/dL).
* The patient has a screening potassium value of >5.5 mmol/L (5.5 mEq/L).
* The patient has a history of alcohol or illicit drug use disorder (as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition).
* The patient has a history of serious side effects or allergic response to any AngII or ERA, including sparsentan, or has a hypersensitivity to any of the excipients in the IMP.
* The female patient is pregnant, plans to become pregnant during the course of the trial, or is breastfeeding.
* The patient has participated in a trial of any investigational product within 28 days prior to screening, or plans to participate in such a trial during the course of this trial.
* The patient, in the opinion of the Investigator, is unable to adhere to the requirements of the trial, including the ability to swallow the IMP whole.
* The patient, in the opinion of the Investigator, has a medical condition or abnormal clinically significant laboratory screening value not listed above that may interfere with the evaluation of sparsentan safety or activity.
* Patients with a medical condition or abnormal clinically significant laboratory screening value not listed above that may interfere with the evaluation of sparsentan safety or activity will be reviewed before consideration of the patient for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Urine protein/creatinine ratio (UP/C) at Week 36 | Week 36
  The primary efficacy endpoint is the change from baseline in the urine protein/creatinine ratio (UP/C), based on a 24-hour urine sample, at Week 36.

SECONDARY OUTCOMES:
eGFR over a 52-week period | Week 58
  Rate of change in eGFR over a 1-year (52 week) period following the initial acute effect of therapy (ie, from 6 weeks post-initiation of investigational medicinal product (IMP) to 58 weeks post-initiation of IMP).
eGFR over a 104-week period | Week 110
  Rate of change in eGFR over a 2-year (104 week) period following the initial acute effect of therapy (ie, from 6 weeks post-initiation of investigational medicinal product (IMP) to 110 weeks post-initiation of IMP).
Change from baseline in proteinuria | Up to Week 114
  Change from baseline in proteinuria, measured by urinary protein/creatinine ratio [UPCR] and 24-hour protein excretion, up to Week 114
Abnormalities in clinical laboratory assessments and vital signs | Up to Week 114
  Proportion of patients with abnormalities in clinical laboratory assessments and vital signs at each visit
Incidence of adverse events (AEs), serious AEs, AEs leading to discontinuation, AEs leading to death | Up to Week 114
  AEs, serious AEs, AEs leading to discontinuation, AEs leading to death

CONTACTS AND LOCATIONS:
Overall Officials: Chee Kay Cheung, MBChB PhD, Principal Investigator — University of Leicester
Locations (5):
- United Kingdom (5):
  - Cambridge University Hospitals NHS Trust, Cambridge, England
  - Northern Care Alliance NHS Foundation Trust - Salford Royal, Salford, England
  - Royal Infirmary of Edinburgh & Western General Hospital, Edinburgh, Scotland
  - University Hospital of wales, Cardiff, Wales
  - Leicester General Hospital, University Hospitals of Leicester NHS Trust, Leicester

IPD SHARING:
Plan to Share IPD: No